CLINICAL TRIAL: NCT06624722
Title: Evaluation of Relationships Between Postural Habits and Awareness With Spine Pain, Spine Functions and Quality of Life in Research Assistant Physicians
Brief Title: Postural Habits, Awareness and Spine
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, doctor, Ufuk University
Other Study IDs: 23.01.12.01/01
Record Dates: First submitted 2024-09-24; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Spine; Posture

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alterations in posture are frequently seen as a risk factor for the development of spine pain. Postural awareness is essential for sustaining healthy postural habits in daily life. The first of the contribution to literature of our study is that the Postural Habits and Awareness Scale, which is a new questionnaire that provides easy inquiry about postural habits and awareness, is a low-cost method and has not been used in the literature before, was used to confirm the relationships between spine pain and functionality and scale parameters in accordance with the literature. Another contribution is that it is underlined that even among doctors, who are the direct managers of health, low postural awareness and bad postural habits that can lead to spinal problems are quite common.

ELIGIBILITY:
Inclusion Criteria:

* participants between the ages of 20-50
* who were working as research assistant physicians

Exclusion Criteria:

* with a history of previous trauma or surgery that could cause pain or postural disorders in the spine,
* known systemic, neurological, psychiatric, infectious, inflammatory, rheumatic, tumoral or degenerative diseases

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 72 volunteer participants between the ages of 20-50 who were working as research assistant physicians.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Postural Habits and Awareness Scale | 1 month
  Postural Habits and Awareness Scale:
  It is a five-point Likert type scale (1=I completely disagree, 5=I completely agree) developed to evaluate postural habits and posture awareness, consisting of 7 items evaluating postural habits and 12 items evaluating postural awareness. In the scale, two main scores are postural habit (PH) and postural awareness (PA); and sub-scores are stance habits and awareness (SHA), awareness of factors that impair stance (AFIS), positional awareness (POA) and ergonomic awareness (EA). Higher scores on the scale indicate better postural habits and awareness levels. The scale was developed by Bayar et al in 2022 and its Turkish validity and reliability study was conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided